CLINICAL TRIAL: NCT07344571
Title: Investigating the Correlation Between Functional Constipation and Sacroiliac Joint Disorders
Acronym: SIJ disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Emad Eldin Mohamed, associate professor, Middle East University
Other Study IDs: 2517
Record Dates: First submitted 2026-01-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Constipation
Keywords: constipation; sacroiliac joint disorders
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Patients with constipation: Both the rectum and the sacroiliac joint share innervation from sacral spinal segments S2-S4. Neural signals from the rectum can influence SI joint sensory nerves via viscerosomatic and somatovisceral reflex arcs. This means chronic constipation may both result from and contribute to SI joint dysfunction.
- group B: Patients without constipation: Accumulated stool in the rectum and sigmoid colon can physically press on pelvic structures, stretching ligaments and tensioning muscles around the SI joint. This may trigger or mimic SI joint dysfunction.

SUMMARY:
Constipation is a common gastrointestinal issue affecting individuals worldwide. Interferential therapy, a form of electrotherapy, has been suggested to have potential benefits in improving gastrointestinal motility and relieving constipation symptoms. Introducing of a new method like electronic cupping therapy with interferential therapy may optimize the therapeutic outcomes by potentially increasing bowel movements and improving overall gastrointestinal function.

DETAILED DESCRIPTION:
Objective: The purpose of this study was to Investigate the correlation between functional constipation and sacroiliac joint disorders Methods: This study involved 200 patients with chronic constipation, consisting of 120 females and 80 males, ranging in age from 25 to 60 years. All participants were allocated into two groups: Group (A) patients with constipation, Group (B) patients without constipation

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* history of Chronic Constipation (CC), as defined by either experiencing two or fewer Complete Spontaneous Bowel Movements (CSBMs) per week for a minimum of 6 consecutive months before the screening visit
* Reporting a sensation of incomplete evacuation or straining during at least a quarter of their bowel movements (according to the generally accepted definition of constipation).
* Patients must have had CC persisting for more than 6 months, failed to respond to or be intolerant of medical treatment for at least 3 months

Inclusion Criteria (for group B):

Not having functional constipation

Exclusion Criteria:

* - pregnant or lactating women
* Chronic Constipation (CC) resulting from anorectal malformations such as colorectal or anal organic lesions, pelvic floor disorders requiring surgical intervention as determined by the investigator (such as rectal prolapse, rectocele, or enterocele)
* presence of implanted electronic devices like cardiac pacemakers, defibrillators, cardiac pumps, or spinal stimulators
* CC attributable to medications or neurologic, endocrine, or metabolic conditions
* prior history of partial colectomy; conditions like megacolon, megarectum, or colonic inertia
* skin abnormalities that hinder the placement of electrodes
* women lacking adequate contraception (hormonal or intrauterine device).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: male and female participant
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Distraction Test (SI Joint Gapping) | 6 months
  Position of patient: Supine. force: posterior-lateral force to both ASISs at same time results: pain in SI region
Thigh Thrust Test | 6 months
  Position of patient: Supine, hip and knee of affected side flexed 90°. force: Stabilize opposite ASIS, apply posterior force through femur. result: Focal SI pain.
Sacral Thrust Test | 6 months
  Position of patient: Prone. force: Apply an anterior shear force to sacrum (over S2). result: Reproduction of pain in SI region.

CONTACTS AND LOCATIONS:
Locations (1):
- Bassam Ahmed Nabil, October City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No